CLINICAL TRIAL: NCT00570570
Title: Muscular Strengthening for Paretic Knee Flexor and Extensor by Conventional Physiotherapy on Chronic Hemiplegic Stroke Patients
Acronym: RenforcHémi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: University Hospital, Bordeaux (Other); University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 07 020 08; PHRC (Other Grant/Funding Number: 07 020 08)
Record Dates: First submitted 2007-12-07; First posted 2007-12-11 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Hemiplegia; Stroke
Keywords: stroke; hemiplegia; gait; Strengthening; Physiotherapy
MeSH Terms: conditions — Hemiplegia; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- group 1 (Other): Muscular Strengthening for paretic knee flexor and extensor
  Interventions: Procedure: Muscular Strengthening for paretic knee flexor and extensor
- group 2 (Active Comparator): conventional physiotherapy
  Interventions: Other: conventional physiotherapy

INTERVENTIONS:
Procedure: Muscular Strengthening for paretic knee flexor and extensor — thrice a week during 6 weeks
  Arms: group 1
Other: conventional physiotherapy — trice a week during 6 weeks
  Arms: group 2

SUMMARY:
Gait impairment remain one of the main problem for hemiplegic stroke patients. After the 6 first months, stroke patients are classically described with moderate or no improvement. Here, we want to compare the effectiveness of a flexor and extensor paretic knee muscular strengthening program with conventional physiotherapy delivered by the local physiotherapist of the patient, in a very ecological way.

DETAILED DESCRIPTION:
Gait impairment remain one of the main problem for most of chronic hemiplegic stroke patients. After the 6 first months, stroke patients are classically described with moderate or no improvement for motor skills. However, physiothertapy is very often delivered to try to increase motor performance. Here, we want to compare the effectiveness of a flexor and extensor paretic knee muscular strengthening program with conventional physiotherapy delivered by the local physiotherapist of the patient, in a very ecological way. Patients will be randomly affected to one group with the same amount of physiotherapy (at least 3 times weekly for 6 weeks). Assessment will be done blindly by another physiotherapist, before, after the 6-week treatment and 6 weeks later to evaluate immediate and remaining benefits of each treatment.

ELIGIBILITY:
Inclusion Criteria:

* Hemipegia due to ischaemic or hemorrhagic stroke more than 6 months ago
* 1st and unique cerebral lesion (Xscan or MRI)
* ability to walk 15 m with or without cane or crutch
* able to understand and give approved consent
* quadriceps at 3/5 (MRC) or stronger

Exclusion Criteria:

* Current treatment with botulinum toxin for spasticity of the paretic flexor or extensor of the knee
* Cardiovascular disease contra-indicating effort and strengthening
* Pregnancy
* Evolving pathology
* Rheumatic disease of the knee contraindicating strengthening
* Aphasia with severe comprehension impairment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2008-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Gait comfortable speed | 3 months

SECONDARY OUTCOMES:
gait analysis (gait maximal speed, kymographic and dynamometric analysis, quality of gait parameter) FIM MOS-SF36 Spasticity (Tardieu Scale) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Xavier D de Boissezon, Principal Investigator — University Hospital, Toulouse
Locations (5):
- France (5):
  - Centre Mutualiste de Rééducation Fonctionnelle, rue Angély Cavlié, Albi
  - Service de Médecine Physique et de Réadaptation, Hôpital Pellegrin, CHU de Bordeaux,, Bordeaux
  - Service de Médecine Physique et de Réadaptation, Hôpital Jean Rebeyrol, CHU de Limoges,, Limoges
  - Service de Médecine Physique et de Réadaptation, Hôpital de Salies du Salat, Salies-du-Salat
  - Service de Médecine Physique et de Réadaptation, Hôpital Rangueil, CHU de Toulouse, TSA 50032, Toulouse